CLINICAL TRIAL: NCT06768983
Title: A Pilot Trial of Strategies to Reduce Fatigue for People With Chronic Kidney Disease (CKD)
Brief Title: Fatigue Reduction in Chronic Kidney Disease (CKD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-01055
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases; Fatigue
MeSH Terms: conditions — Renal Insufficiency, Chronic; Fatigue | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remotely Delivered Cognitive Behavioral Therapy (CBT) (Experimental): Patients with non-dialysis dependent kidney disease who have complaints of fatigue will be enrolled. Participants will receive remotely delivered CBT sessions, which will weekly with the goal of having 10 45-minute sessions over 12 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — 10 sessions of remotely delivered CBT; each session is about 45 minutes in length. The aim of the sessions is to cultivate skills that promote activity and reduce fatigue and its impact on daily activities.

SUMMARY:
In this pilot trial, investigators will pilot test a cognitive behavioral intervention for acceptability and proof of concept for a larger future trial to be submitted for federal funding. This is a one-group design with qualitative and quantitative data collection integrated into the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Interest in participating in a fatigue study
* Age ≥18 years old
* Estimated glomerular filtration rate (eGFR) 15-44 mL/min/1.73 m2
* Ability and willingness to provide informed consent
* Ability to speak English
* Ability to walk
* Ability to join remote study sessions via WebEx

Exclusion Criteria:

* Current involvement in an activity/exercise program
* High likelihood of a kidney transplant within 6 months (assessed via the medical record)
* Any safety concerns about increased walking (assessed via the medical record)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Session Adherence | Up to Week 12
  Measure of feasibility; calculated as the percentage of planned sessions that were actually attended by participants.

SECONDARY OUTCOMES:
Change in Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Score | Baseline, Week 6
  The FACIT Measurement System is a collection of health-related quality of life (HRQOL) questionnaires targeted to the management of chronic illness. The Fatigue Subscale comprises 13 items and measures symptoms of fatigue. Each item is rated on a scale from 0 (not at all) to 4 (very much); the total score is the sum of responses and ranges from from 0 to 52; lower scores indicate greater fatigue.
Change in Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Score | Baseline, Week 12
  The FACIT Measurement System is a collection of health-related quality of life (HRQOL) questionnaires targeted to the management of chronic illness. The Fatigue Subscale comprises 13 items and measures symptoms of fatigue. Each item is rated on a scale from 0 (not at all) to 4 (very much); the total score is the sum of responses and ranges from from 0 to 52; lower scores indicate greater fatigue.
Change in Dialysis Symptom Index (DSI) Score | Baseline, Week 6
  The DSI is 30-item assessment of CKD-related unpleasant symptoms. Each item is rated on a scale from 0 (not at all) to 4 (very much). The total score is the sum of the responses, ranging from 0 to 120. A higher score indicates a greater symptom burden.
Change in Dialysis Symptom Index (DSI) Score | Baseline, Week 12
  The DSI is 30-item assessment of CKD-related unpleasant symptoms. Each item is rated on a scale from 0 (not at all) to 4 (very much). The total score is the sum of the responses, ranging from 0 to 120. A higher score indicates a greater symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cukor, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Daniel.Cukor@nyulangone.org. The protocol will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Daniel.Cukor@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.